CLINICAL TRIAL: NCT01392339
Title: Sleep Apnea: Interface Between Basic and Clinical Research
Brief Title: Obstructive Sleep Apnea and Genes Expression
Acronym: HIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associacao Fundo de Incentivo a Psicofarmcologia (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Lia Rita Azeredo Bittencourt, Associacao Fundo de Incentivo a Psicofarmacologia - AFIP
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 0985/08
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; CPAP; hypoxia; sleep; translational science; gene expression
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypoxia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CPAP (Experimental): CPAP - Continuous Positive Airway Pressure, gold standard treatment to Obstructive Sleep Apnea
  Interventions: Procedure: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Procedure: Continuous Positive Airway Pressure (CPAP) — Continuous Positive Airway Pressure (CPAP) is a method of respiratory ventilation used primarily in the treatment of obstructive sleep apnea

SUMMARY:
Obstructive sleep apnea is a multi-component disease. This study will test the hypotheses that hypoxia per se modulates gene expression in animal model of sleep apnea and these results may be translated with alterations that occur in apneic patients. Thus, we aim to integrate basic and clinical research to shed light on novel candidate genes involved in sleep apnea.

DETAILED DESCRIPTION:
Twenty-four male rats were exposed to chronic intermittent hypoxia (5% O2) or normoxia for 6 wks. Following chronic intermittent hypoxia, a group of 8 rats were removed from the chronic intermittent hypoxia protocol and allowed to normoxic conditions over a period of 2 wks. For the clinical protocol, the AHI measured by overnight polysomnography will be use to select individuals with sleep-related breathing disorders, and controls (30-60 years, Body Mass Index (BMI) < 35kg/m2). Moreover, the investigators will evaluate the subjective sleep parameters (sleep disorders questionnaire, the Epworth Sleepiness Scale, sleep diaries). After standard CPAP titration, men with severe obstructive sleep apnea will be assigned for the CPAP protocol for future assessment of the influence of 6 months obstructive sleep apnea treatment. A total of 84 genes are evaluated using the Hypoxia Signaling Pathway PCR Array (SA Biosciences, EUA).

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged between 30 and 60 years old
* Normal range of laboratory tests complete blood count (CBC), glucose, total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL) and very low-density lipoprotein (LDL), triglycerides
* Body Mass Index (BMI) < 35kg/m2

Exclusion Criteria:

* Presence of clinical diseases (chronic obstructive pulmonary disease, asthma, interstitial lung diseases, neuromuscular diseases, heart failure, thyroid disease, rheumatologic and psychiatric) and other sleep disorders
* Smoking status
* Participants who had current or historical treatment with CPAP or any other treatment for OSA
* Presence of anatomical obstructive upper airway, tonsil grade III and IV septal deviation and grade III (severe) that may affect the outcome of CPAP
* Alcoholism
* Use of sleep-inducing medications

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Apnea/Hypopnea Index | 6 months after the basal evaluation
  Polysomnographic date of sleep stages percentages, sleep efficiency, arousals, apnea-hypopnea index, oxyhemoglobin saturation

SECONDARY OUTCOMES:
Gene expression | 6 months after the basal evaluation
  A total of 84 genes are evaluated using the Hypoxia Signaling Pathway PCR Array (SA Biosciences, EUA), C-reactive protein (CRP), and biochemical parameters

CONTACTS AND LOCATIONS:
Overall Officials: Juliana C Perry, PhD, Principal Investigator — Federal University of São Paulo; Lia Rita A Bittencourt, MD, PhD, Study Director — Associacao Fundo de Incentivo a Psicofarmacologia
Locations (1):
- AFIP - Instituto do Sono (Sleep Institute), São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Hypoxia Signaling Pathway PCR Array (SA Biosciences, EUA) — http://www.sabiosciences.com/
- See also: American Academy of Sleep Medicine — http://www.aasmnet.org/